CLINICAL TRIAL: NCT01864564
Title: Early Gestational Diabetes Screening in the Gravid Obese Woman
Acronym: EGGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Ochsner Health System (Other)
Responsible Party: Principal Investigator, Lorie M Harper, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: F121008004; K12HD001258 (NIH)
Record Dates: First submitted 2013-05-22; First posted 2013-05-29 (Estimated); Results first posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Gestational Diabetes; Obesity
Keywords: Gestational diabetes; Screening; Obesity; Anhydroglucitol
MeSH Terms: conditions — Diabetes, Gestational; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine Screening (No Intervention): Obese women will be screened at 24-28 weeks of gestation for gestational diabetes using the standard U.S. screening method of a 1-hour, 50-g glucose challenge test followed by a 3-hour, 100-g glucose tolerance test if abnormal. Women identified as having diabetes will be treated according to standards of care.
  All women will have a hemoglobin A1c and 1,5-anhydroglucitol checked at 14-18 weeks and 24-28 weeks gestation.
- Early Screening (Experimental): Obese women will be randomized to be screened at 14-19.9 weeks of gestation for gestational diabetes using the standard U.S. screening method of a 1-hour, 50-g glucose challenge test followed by a 3-hour, 100-g glucose tolerance test if abnormal. Women identified as having diabetes will be treated according to standards of care. Women who do not have diabetes at 14-19.9 weeks will be re-screened at 24-28 weeks per the standard of care.
  All women will have a hemoglobin A1c and 1,5-anhydroglucitol checked at 14-18 weeks and 24-28 weeks gestation.
  Interventions: Other: Early Screen

INTERVENTIONS:
Other: Early Screen — Women will be randomized to be screened for gestational diabetes at 14-19.9 weeks gestation (early=intervention) versus routine screening at 24-28 weeks.
  Arms: Early Screening

SUMMARY:
Specific Aim 1: To test the hypothesis that early GDM screening between 14-18 weeks in obese women (body mass index ≥30.0) will result in improved perinatal outcomes.

Specific Aim 2: To test the hypothesis that a lower diagnostic threshold for GDM at 14-18 weeks will result in improved detection of GDM and reduce the need for third-trimester testing.

Specific Aim 3: To test the hypothesis that 1,5-anhydroglucitol, a sensitive marker of hyperglycemia, can be used as a simple and sensitive serum test for GDM in the obese population.

DETAILED DESCRIPTION:
Over 1/3 of reproductive age women are obese. Obese women have higher rates of adverse pregnancy outcomes, including stillbirth, fetal growth disorders, diabetes, hypertensive diseases and maternal death. Although weight loss prior to pregnancy is the ideal, a significant proportion of obese women do not present to care until after conception. Consequently, developing a comprehensive plan for managing the obese gravida is imperative. One component of such a plan must include screening and treating for gestational diabetes (GDM), which is associated with macrosomia, cesarean delivery, preeclampsia, shoulder dystocia, and neonatal hypoglycemia. Obesity substantially increases the risk of GDM (odds ratio 2-5). GDM treatment has been shown to improve pregnancy outcomes,but obese women with GDM continue to have worsened outcomes compared to normal weight women with GDM, with more cesarean delivery, preeclampsia, macrosomia and stillbirths occurring in obese women. This is perhaps due to pre-existing insulin resistance in obese women that, when coupled with the normal insulin resistance of pregnancy, leads to earlier onset of GDM in obese women compared to normal weight women, with consequently longer fetal exposure to hyperglycemic episodes prior to diagnosis and treatment.

The American College of Obstetricians and Gynecologists recommends screening obese women for gestational diabetes (GDM) in the first trimester or upon presentation. However, due to lack of supporting data, this recommendation is not widely followed and the majority of obese women do not undergo GDM screening until 24-28 weeks gestation. Postponing testing may delay the diagnosis and treatment of GDM by 10 weeks or more, resulting in fetal hyperglycemia during critical periods of fetal growth and development. Early screening, between 14-18 weeks gestation, in this high-risk population will allow for earlier recognition and treatment of GDM, thereby improving perinatal outcomes.

Additionally, little is known about screening and diagnostic standards for GDM early in pregnancy. Currently, when GDM testing is performed early in pregnancy, the criteria used to diagnose GDM at 24-28 weeks are applied. However, these thresholds were developed for a test performed at 24-28 weeks; applying these same thresholds at 14-18 weeks may not be appropriate. As insulin resistance increases throughout pregnancy, lowering the criteria for glucose tolerance testing earlier in gestation may improve GDM detection and avoid the need for re-testing later in pregnancy. Alternatively, as GDM is the new-onset of insulin resistance with resulting hyperglycemia, biomarkers that reflect metabolic markers of recent hyperglycemic episodes may perform well in screening for GDM and may decrease the patient burden of, while increasing compliance with, glucose tolerance testing. One such marker that has been evaluated in Type 2 diabetes is 1,5-anhydroglucitol (AG), an unmetabolized monosaccharide. AG has a fairly stable steady-state concentration in the blood that is unaffected by fasting, dietary changes and pregnancy; it is reabsorbed in the renal tubules by the same transporter that reabsorbs glucose. During a hyperglycemic episode, the presence of glucose in the urine competitively inhibits the reabsorption of AG, resulting in a precipitous decline in AG levels. AG levels recover slowly in the presence of continued hyperglycemia. The rapid fall of AG with the onset of hyperglycemia and its slow recovery in situations of on-going hyperglycemia suggest it as both a sensitive and specific marker for new-onset glucose intolerance requiring treatment. As perinatal outcomes are closely linked to hyperglycemic excursions, (18) AG may be the most sensitive and specific marker for determining the GDM patient who will benefit most from treatment.

This study is potentially practice changing and could greatly reduce the disparities in perinatal outcomes seen in obese women. Early GDM screening of obese women may reduce the risk of cesarean delivery, macrosomia, stillbirth, preterm birth, and preeclampsia in this population. This study has 3 specific aims:

Specific Aim 1: To test the hypothesis that early GDM screening between 14-18 weeks in obese women (body mass index ≥30.0) will result in improved composite perinatal outcomes.

Specific Aim 2: To test the hypothesis that a lower diagnostic threshold for GDM at 14-18 weeks will result in improved detection of GDM and reduce the need for third-trimester testing.

Specific Aim 3: To test the hypothesis that 1,5-anhydroglucitol, a sensitive marker of recent hyperglycemic excursions, can be used as a simple and sensitive serum test for GDM in the obese population.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* 18 years and older
* Body mass index >=30.0
* <20 weeks gestation at presentation for care

Exclusion Criteria:

* Prior cesarean
* History of bariatric surgery
* Major maternal medical illness (cardiac disease, HIV, hemoglobinopathy, oxygen requirement)
* Chronic prednisone use
* Known fetal anomalies
* Multifetal gestation

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 962 (Actual)
Dates: Start 2013-06-18 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorie M Harper, MD, MSCI, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Ochsner Health System, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harper LM, Jauk V, Longo S, Biggio JR, Szychowski JM, Tita AT. Early gestational diabetes screening in obese women: a randomized controlled trial. Am J Obstet Gynecol. 2020 May;222(5):495.e1-495.e8. doi: 10.1016/j.ajog.2019.12.021. Epub 2020 Jan 9. PMID 31926951

RESULTS

PARTICIPANT FLOW:
Groups:
- Early Screening: Obese women will be randomized to be screened at 14-19.9 weeks of gestation for gestational diabetes using the standard U.S. screening method of a 1-hour, 50-g glucose challenge test followed by a 3-hour, 100-g glucose tolerance test if abnormal. Women identified as having diabetes will be treated according to standards of care. Women who do not have diabetes at 14-19.9 weeks will be re-screened at 24-28 weeks per the standard of care.
  All women will have a hemoglobin A1c and 1,5-anhydroglucitol checked at 14-18 weeks and 24-28 weeks gestation.
  Early Screen: Women will be randomized to be screened for gestational diabetes at 14-19.9 weeks gestation (early=intervention) versus routine screening at 24-28 weeks.
Period: Overall Study
Arm/Group | Routine Screening | Early Screening
Started | 480 | 482
Completed | 443 | 387
Not Completed | 37 | 95
Not completed — Lost to Follow-up | 17 | 23
Not completed — Withdrawal by Subject | 20 | 11
Not completed — Protocol Violation | 0 | 27
Not completed — not reported | 0 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Routine Screening | Early Screening | Total
Number analyzed (Participants) | 463 | 459 | 922
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.8 (5.9) | 27.2 (5.9) | 27 (5.9)
Sex/Gender, Customized [Count of Participants; unit: Participants] — All participants were female
  Participants
    female | 463 | 459 | 922
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, Non-Hispanic | 35 | 52 | 87
  Black, Non-Hispanic | 299 | 280 | 579
  Native American | 3 | 2 | 5
  Asian | 2 | 1 | 3
  Hispanic | 123 | 122 | 245
  Other | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 463 | 459 | 922
Region of Enrollment [Number; unit: participants]
  United States | 463 | 459 | 922
Body Mass index at randomization [Mean (Standard Deviation); unit: kg/m^2] | 37.0 (6.5) | 37.2 (6.6) | 37 (0.6)
Medicaid/no insurance [Count of Participants; unit: Participants] | 441 | 434 | 875
Married [Count of Participants; unit: Participants] | 96 | 98 | 194
High School education or greater [Count of Participants; unit: Participants] | 305 | 309 | 614
Parous [Count of Participants; unit: Participants] | 338 | 329 | 667
Any Smoking [Count of Participants; unit: Participants] | 98 | 83 | 181
Any alcohol use [Count of Participants; unit: Participants] | 61 | 76 | 137
Any drug use [Count of Participants; unit: Participants] | 49 | 41 | 90
Hypertension [Count of Participants; unit: Participants] | 50 | 61 | 111
Asthma [Count of Participants; unit: Participants] | 53 | 61 | 114
Depression [Count of Participants; unit: Participants] | 50 | 55 | 105
Hemoglobin A1c at 14-20 weeks [Mean (Full Range); unit: % A1c] | 5.3 [5.0 to 5.6] | 5.3 [5.0 to 5.6] | 5.3 [5.0 to 5.6]
Gestational age at Randomization [Mean (Standard Deviation); unit: weeks] | 13.6 (3.7) | 13.8 (3.8) | 13.7 (3.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Composite Perinatal Outcome
Description: Any one of the following: Macrosomia (birth weight > 4000 g), primary cesarean, gestational hypertension, preeclampsia, shoulder dystocia, neonatal hyperbilirubinemia, neonatal hypoglycemia (<40 mg/dL)
Time Frame: Baseline to within 6 weeks of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Screening | Early Screening
Number analyzed (Participants) | 463 | 459
Participants | 235 | 261

2. Secondary Outcome: Number of Participants With Macrosomia
Description: Number of infants with Birth weight >4000 g
Time Frame: Within 6 weeks of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Screening | Early Screening
Number analyzed (Participants) | 463 | 459
Participants | 21 | 25

3. Secondary Outcome: Primary Cesarean Delivery
Description: Primary cesarean : delivery via cesarean, first cesarean (does not include repeat cesarean deliveries)
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Screening | Early Screening
Number analyzed (Participants) | 463 | 459
Participants | 93 | 79

4. Secondary Outcome: Pregnancy Induced Hypertension
Description: Includes gestational hypertension and preeclampsia
Time Frame: Within 6 weeks of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Screening | Early Screening
Number analyzed (Participants) | 463 | 459
Participants | 102 | 136

5. Secondary Outcome: Shoulder Dystocia
Description: Shoulder dystocia as identified by delivering physician
Time Frame: At birth
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Screening | Early Screening
Number analyzed (Participants) | 463 | 459
Participants | 32 | 30

6. Secondary Outcome: Neonatal Hyperbilirubinemia
Description: serum bilirubin level above the 95th percentile for gestational age
Time Frame: Within 6 weeks of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Screening | Early Screening
Number analyzed (Participants) | 463 | 459
Participants | 72 | 90

7. Secondary Outcome: Neonatal Hypoglycemia
Description: Blood sugar level <40 mg/dL
Time Frame: Within 6 weeks of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Screening | Early Screening
Number analyzed (Participants) | 463 | 459
Participants | 19 | 22

8. Secondary Outcome: Gestational Age at Delivery
Description: Gestational age in weeks as calculated by ACOG criteria
Time Frame: at delivery
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Routine Screening | Early Screening
Number analyzed (Participants) | 463 | 459
weeks | 38.5 (3.4) | 38.2 (4.4)

9. Secondary Outcome: Any Diabetic Medication
Description: includes the use of any diabetic medication
Time Frame: baseline to delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Screening | Early Screening
Number analyzed (Participants) | 463 | 459
Participants | 20 | 31

10. Secondary Outcome: Insulin Medication
Description: Includes the use of Insulin
Time Frame: baseline to delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Screening | Early Screening
Number analyzed (Participants) | 463 | 459
Participants | 3 | 11

11. Secondary Outcome: Large for Gestational Age
Description: defined as >= the 90th percentile by Duryea et al
Time Frame: at delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Screening | Early Screening
Number analyzed (Participants) | 463 | 459
Participants | 26 | 27

ADVERSE EVENTS:
Time Frame: Baseline through 8 months
Arm/Group | Routine Screening | Early Screening
All-Cause Mortality (participants affected / at risk) | 10/463 | 22/459
Serious Adverse Events (participants affected / at risk) | 10/463 | 22/459
Other Adverse Events (participants affected / at risk) | 1/463 | 0/459
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Routine Screening (N=463) | Early Screening (N=459)
Fetal or Neonatal death (Pregnancy, puerperium and perinatal conditions) | 10 (10) | 22 (22)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Routine Screening (N=463) | Early Screening (N=459)
Other - Preterm Delivery (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — Preterm delivery

LIMITATIONS AND CAVEATS:
Lack of blinding of participants and providers may have introduced bias. The study population being largely Black or Hispanic women and without private insurance limits the generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-03-29): https://cdn.clinicaltrials.gov/large-docs/64/NCT01864564/SAP_000.pdf
  • Study Protocol (2014-02-17): https://cdn.clinicaltrials.gov/large-docs/64/NCT01864564/Prot_001.pdf